CLINICAL TRIAL: NCT03371095
Title: Multicenter, Randomized, Prospective Trial Comparing the Efficacy and Safety of Infliximab to That of Cyclophosphamide in Severe Behçet's Disease. ITAC : Induction Therapy With Anti-TNFα vs Cyclophosphamide in Severe Behçet Disease
Brief Title: Induction Therapy With Anti-TNFα vs Cyclophosphamide in Severe Behçet Disease
Acronym: ITAC
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P160932J
Record Dates: First submitted 2017-12-07; First posted 2017-12-13 (Actual); Last update posted 2023-07-03 (Actual); Status verified 2017-12

CONDITIONS: Behcet's Disease; Vasculitis
Keywords: Behcet's Disease; Vasculitis; Biotherapy; immunosuppressant; Infliximab
MeSH Terms: conditions — Behcet Syndrome; Vasculitis | interventions — Infliximab; Cyclophosphamide

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Infliximab (Experimental): Infliximab 5mg/kg intravenously at week 0, 2, 6, 12, and 18
  Interventions: Drug: Infliximab
- Cyclophosphamide (Active Comparator): Cyclophosphamide 0.7g/m2 up to 1.2g/m2 intravenously at week 0, 4, 8, 12, 16 and 20
  Interventions: Drug: Cyclophosphamide

INTERVENTIONS:
Drug: Infliximab — Use of infliximab instead of cyclophosphamide
  Arms: Infliximab
Drug: Cyclophosphamide — Use of cyclophosphamide
  Arms: Cyclophosphamide

SUMMARY:
Behçet's disease (BD) is a systemic vasculitis of arterial and venous vessels of any size, involving young patients (from 15 to 45 years). BD significantly increases morbidity and mortality. Therapeutic management of BD depends on the clinical presentation and organ involved. Although colchicine, nonsteroidal antiinflammatory agents and topical treatments are often sufficient for mucocutaneous and joint involvement, more aggressive approach with immunosuppressive agents is warranted for severe manifestations. Early recognition and vigorous use of immunosuppressives with high dose steroids have changed the prognosis of patients with severe BD. BD is a severe systemic vasculitis leading to blindness in up to 20% at 4 years and a 5-year mortality rate of 15% in patients with major vessel or neurological involvement. Cyclophosphamide has been used for life-threatening BD for 40 years. However, the outcome of severe complications of BD is poor. The European League Against Rheumatism (EULAR) recommendation for the management of BD advocated cyclophosphamide plus glucocorticoids for life-threatening manifestations (i.e neurological and/or major vessel involvement). TNFa antagonists have been used with success in severe and/or resistant cases. In addition, the incidence of blindness in BD has been dramatically reduced in the recent years with the use of anti-TNF. However, there is no firm evidence or randomized controlled trials directly addressing the best induction immunosuppressive therapy in severe BD manifestations. The investigators therefore aimed to assess the best induction therapy in severe and difficult to treat BD patients. The investigators hypothesize that up to 70% of the patients with life-threatening manifestations of BD receiving these compounds [anti-TNFa or cyclophosphamide] will achieve a complete remission of BD at 6 months and with less than 0.1 mg/kg/day of prednisone.

ITAC, is the first randomized prospective, head to head study, comparing infliximab, to cyclophosphamide in severe manifestations of BD. There is no firm evidence or randomized controlled trials directly addressing the best induction immunosuppressive therapy in severe BD. Cyclophosphamide failed to demonstrate sustainable remission over 70 % of life threatening BD cases. There is little published information on use of immunosuppressants other than cyclophosphamide for severe BD. TNFa antagonists have been used with success in severe and/or resistant cases. TNFa expression correlates with BD activity and other immunological data provide a strong rationale for targeting BD with biologics. Despite a strong rationale, these compounds are not yet approved in BD, which guarantees the innovative nature of this study that aims selecting or dropping any arm when evidence of efficacy already exists.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 12 years old
* Written inform consent (Informed Consent should be obtained from the legal guardian in accordance with regional laws or regulations for patients 12 to 17 years of age)
* Diagnosis of BD according to international criteria for BD (ICBD) (see Appendix 1).
* Life threatening active BD defined as 1 of the following disease categories and according to the validated international definition:

  * Major vessel disease: arterial aneurysms or arterial stenosis, myocarditis and/or major deep vein thrombosis (i.e. inferior vena cava, superior vena cava, cardiac cavity thrombosis, pulmonary embolism, supra-hepatic vessels, renal and mesenteric vessels). Diagnosis of major vessel involvement will be done using vascular doppler sonography, echocardiography, angio-CT scan and/or cardiac magnetic resonance imaging (MRI).
  * Central nervous system involvement: encephalitis or meningoencephalitis or myelitis. The diagnosis of neuro-Behçet's (CNS involvement) will be based on objective neurological symptoms that were associated with neuroimaging (CNS and/or medullar MRI) findings suggestive of BD-related CNS involvement. Cerebrospinal fluid (CSF) findings showing aseptic inflammation may be associated.
* Chest X-ray results (postero-anterior and lateral) within 12 weeks prior to inclusion with no evidence of active Tuberculosis, active infection, or malignancy
* For female subjects of child-bearing age, a negative pregnancy test
* For subjects with reproductive potential, a willingness to use contraceptive measures adequate to prevent the subject or the subject's partner from becoming pregnant during the study and 6 months after stopping therapy. Adequate contraceptive measures include hormonal methods used for two or more cycles prior to Inclusion (e.g., oral contraceptive pills, contraceptive patch, or contraceptive vaginal ring), barrier methods (e.g., contraceptive sponge, diaphragm used in conjunction with contraceptive foam or jelly, or condom used in conjunction with contraceptive foam or jelly), intrauterine methods (IUD), sterilization (e.g., tubal ligation or a monogamous relationship with a vasectomized partner), and abstinence.
* A potential subject with a positive interferon-gamma release assay (IGRA) (e.g., QuantiFERON®-TB Gold or T-spot TB® Test) or a positive tuberculin skin test (≤6 months) is eligible if her/his chest X-ray does not show evidence suggestive of active tuberculosis (TB) disease and there are no clinical signs and symptoms of pulmonary and/or extra-pulmonary TB disease. These subjects with a latent TB infection who have not already received a prophylactic TB treatment must agree in advance to complete such a treatment course.
* HIV negative serology and negative HBs Ag test (≤1 month)

Exclusion Criteria:

* Evidence of active Tuberculosis
* HIV or active HBV infection (HBs Ag+).
* Pregnancy or lactation
* Have been taking an oral daily dose of a glucocorticoid of more than 20 mg prednisone equivalent for more than 6 weeks continuously prior to the inclusion visit or taking more than 3000 mg methylprednisolone 4 weeks prior to the inclusion visit
* Alcohol or drug dependance
* Severe renal (creatinine clearance <30ml/min/1,73m2) or pre-existing hemorrhagic cystitis or liver insufficiency (hepatic encephalopathy) or urinary obstruction
* Heart failure ≥ stage III / IV NYHA,
* History of malignancy within 5 years prior to Inclusion other than carcinoma in situ of the cervix or excised basal cell or squamous cell carcinoma of the skin.
* History of multiple sclerosis and/or demyelinating disorder
* History of severe allergic or anaphylactic reactions to cyclophosphamide or infliximab
* Infectious disease:

  * Infection requiring treatment with intravenous antibiotics within 2 weeks prior to Inclusion
  * History of recurrent infection
* Laboratory values assessed during Inclusion:

  * Hemoglobin < 8 g/dL
  * WBC < 2.0 x 103/mm3
  * Platelet count < 70 x 103/mm3
* Use of the following systemic treatments during the specified periods:

  * Treatment with systemic biologic therapy or with cyclophosphamide within 3 months prior to Inclusion
  * if on azathioprine, mycophenolate mofetil, or methotrexate at the time of inclusion, these drugs must be withdrawn prior to receiving the cyclophosphamide or infliximab dose on Day 1
* Any live (attenuated) vaccine within 4 weeks prior inclusion; recombinant or killed virus vaccines are permitted.
* Lack of affiliation to a social security benefit plan (as a beneficiary or assignee), patients affiliated to universal medical coverage (CMU) are eligible for the study

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2018-05-25 (Actual); Primary Completion 2021-12-24 (Actual); Study Completion 2022-04-11 (Actual)

PRIMARY OUTCOMES:
Complete clinical response | At week 22 after randomization
  The complete clinical response is defined by the remission of all affected organs involved at baseline with a prednisone ≤ 0.1mg/kg per day

SECONDARY OUTCOMES:
Complete clinical response | At week 12 after randomization
  The complete clinical response is defined by the remission of all affected organs involved at baseline with a prednisone ≤ 0.1mg/kg per day
Complete clinical response | At week 48 after randomization
  The complete clinical response is defined by the remission of all affected organs involved at baseline with a prednisone ≤ 0.1mg/kg per day
Remission of CNS and/or cardiovascular involvement | At week 12 after randomization
Remission of CNS and/or cardiovascular involvement | At week 22 after randomization
Remission of CNS and/or cardiovascular involvement | At week 48 after randomization
Percent meeting the target of ≤ 0.1 mg/day/kg of prednisone | At week 22 after randomization
Percent meeting the target of ≤ 0.1 mg/day/kg of prednisone | At week 48 after randomization
Mean dose of prednisone | At week 12 after randomization
Mean dose of prednisone | At week 22 after randomization
Mean dose of prednisone | At week 48 after randomization
Cumulative dose of prednisone | At week 12 after randomization
Cumulative dose of prednisone | At week 22 after randomization
Cumulative dose of prednisone | At week 48 after randomization
Time to response onset | At week 48 after randomization
C-reactive protein | Every 4 weeks
  CRP in blood sample
Time to relapse | At week 48 after randomization
  Relapse will be defined as the reappearance of clinical and/or paraclinical features of active disease or by the occurrence of new lesions at week 48
Rate of relapse | At week 48 after randomization
Time to occurrence of worsening | At week 48 after randomization
  Worsening will be defined as the progression of preexisting lesions) at week 22 and 48
Rate of worsening | At week 48 after randomization
Overall survival | At week 22 after randomization
Overall survival | At week 48 after randomization
Event Free Survival | At week 22 after randomization
Event Free Survival | At week 48 after randomization
Frequency of adverse clinical events | At week 22 after randomization
  Incidence of Treatment related Adverse Events
Severity of adverse clinical events | At week 22 after randomization
Change in quality of life | At week 12 after randomization
  Change in quality of life (QOL) (SF-36V2TM Health Survey)
Change in quality of life | At week 22 after randomization
  Change in quality of life (QOL) (SF-36V2TM Health Survey)
Changes in CNS involvement | At week 12 after randomization
  Changes in CNS involvement on physical exam, and cerebral and/or medullar MRI.
Changes in CNS involvement | At week 22 after randomization
  Changes in CNS involvement on physical exam, and cerebral and/or medullar MRI.
Changes in vascular involvement | At week 12 after randomization
  Changes in vascular involvement on physical exam, vascular Doppler US, and angio-CT imaging and biologically (normalization of C reactive protein)
Changes in vascular involvement | At week 22 after randomization
  Changes in vascular involvement on physical exam, vascular Doppler US, and angio-CT imaging and biologically (normalization of C reactive protein)
Changes in cardiological involvement | At week 12 after randomization
  Changes in cardiological involvement on physical exam, echocardiography (normalization of left ventricular function and/or disappearance of cardiac thrombosis), and cardiac magnetic resonance imaging (disappearance of gadolinium enhancement and normalization of left ventricular function) and biologically (normalization of troponin and of C reactive protein)
Changes in cardiological involvement | At week 22 after randomization
  Changes in cardiological involvement on physical exam, echocardiography (normalization of left ventricular function and/or disappearance of cardiac thrombosis), and cardiac magnetic resonance imaging (disappearance of gadolinium enhancement and normalization of left ventricular function) and biologically (normalization of troponin and of C reactive protein)
Serum concentration measurement of TNFa inhibitor at week 22 | At week 12 after randomization
Change in Behcet's Disease Current Activity Form | At week 12 after randomization
Change in Behcet's Disease Current Activity Form | At week 22 after randomization

CONTACTS AND LOCATIONS:
Locations (27):
- France (27):
  - CHRU Amiens, Amiens
  - Hôpital Avicenne, Bobigny
  - CHU Bordeaux, Bordeaux
  - Hôpital Saint André, Bordeaux
  - CH Ambroise Paré, Boulogne-Billancourt
  - CHU Caen, Caen
  - Henri Mondor Hospital, Créteil
  - CHU Dijon, Dijon
  - CHU Grenoble, Grenoble
  - CHU Bicêtre, Le Kremlin-Bicêtre
  - CHRU Lille, Lille
  - Hôpital de la Croix Rousse, Lyon
  - Hôpital Edouard Herriot, Lyon
  - Hôpital de La Timone, Marseille
  - CH Metz, Metz
  - CHU Bichat, Paris
  - CHU Tenon, Paris
  - Hôpital de La Pitié Salpetriere, Paris
  - Hôpital Foch, Paris
  - Hôpital Lariboisière, Paris
  - Hôpital Saint Antoine, Paris
  - Hôpital Saint Louis, Paris
  - CHU Poitiers, Poitiers
  - Hôpital Bois Guillaume, Rouen
  - CH Saint-Denis, Saint-Denis
  - CHU Purpan, Toulouse
  - CH Valenciennes, Valenciennes

IPD SHARING:
Plan to Share IPD: Undecided